CLINICAL TRIAL: NCT07155616
Title: Computational Tool for Measuring Arterial Flow From CT
Brief Title: NON-INVASIVE BLOOD FLOW ASSESSMENT: Computational Tool for Measuring Arterial Flow From CT
Acronym: NOVELLA
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: HCB/2023/0531
Record Dates: First submitted 2025-08-12; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Vascular; Surgical Planning
Keywords: surgical planning; pancreatic surgery
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood flow measurement — Intraoperative blood flow measurement

SUMMARY:
Major invasive surgery, such as oncological abdominal surgery, is associated with a high risk of complications and mortality.

One of the main problems in this type of surgery is the difficulty in preserving the arteries and veins necessary to support vital organs.

The main objective of this project is to develop software to predict vascular flow changes based on preoperative computed tomography (CT) scans.

Currently, the only way to assess preoperative vascular flow is through percutaneous angiography. This is an invasive procedure that requires anaesthesia, hospitalisation, high doses of radiation, vessel manipulation and the possibility of serious injury. It is often used for the diagnosis of vascular stenosis, analysis of vascular flow and preoperative planning to determine which vessels are directly related to organ perfusion.

This preoperative planning will be key in the following clinical scenarios:

1. Anomalous hepatic artery anatomy in pancreaticoduodenectomy.
2. Celiac trunk stenosis.
3. Hepatic artery revascularisation from the superior mesenteric artery.
4. Hepatic artery flow assessment in liver transplantation.
5. Splenic artery flow steal phenomenon in liver transplantation.

Novella aims to develop a tool that has the capability to predict postoperative vascular flow.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for pancreaticoduodenectomy.
* Good quality preoperative DICOM CT (arterial phase).
* Michel's I arterial configuration.
* Any surgical approach (open or robotic).
* Informed consent.

Exclusion Criteria:

* Age < 18 years.
* Technical inability to measure flow.
* GDA infiltration.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing pancreaticoduodenectomy for any reason.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy of blood flow modification prediction | 10 months
  Compare software's blood flow modification prediction with introperative measurement in each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided